CLINICAL TRIAL: NCT05192577
Title: Nerve Excitability Testing Protocol for Cold-sensing Fibers
Brief Title: Testing Protocol for Cold-sensing Fibers
Acronym: Cold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Jenny Tigerholm, Assistant Professor, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N-20200014 5-subproject
Record Dates: First submitted 2021-11-23; First posted 2022-01-14 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental)
  Interventions: Other: Electrical stimulation

INTERVENTIONS:
Other: Electrical stimulation — At the beginning of the session, an electrode will be attached to the participant's ankle. Electrical stimulation will be applied to estimate the electrical perception threshold. This threshold will be used as condition stimuli when different thermal thresholds are assessed.

SUMMARY:
This project aims to evaluate whether electrical stimulation can modulate the cold detection threshold and the cold pain threshold. The hypothesis is that different electrical stimulation will either decrease or increase the cold threshold depending on the shape of the electrical stimulus. If a combination of electrical stimuli and cold stimuli could be used, this could lead to a novel method for estimating the excitability properties of cold-sensing fibers. The sub-project takes place in 1 session (1.5 hours).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-80 years
* Speak and understand English

Exclusion Criteria:

* Pregnancy or breast feeding
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Previous and present neurologic, musculoskeletal or mental illnesses (e.g., epilepsy, neuropathy, fibromyalgia and depression)
* Skin diseases
* Past history of conditions possibly leading to neuropathy
* Inability to cooperate
* Current use of medications that may affect the study, e.g., analgesics
* Previous traumatic experience of an electrical accident
* Consumption of alcohol or painkillers within the last 24 hours
* Participation in other pain studies throughout the study period
* Patients with cardiac diseases (e.g., pacemaker).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Cold detection threshold | During session 1. The estimation of the outcome measurement take approximately 3 minutes.
  The cold detection threshold will be estimated by reducing the temperature until the subjects perceive a cold sensation.
Cold detection threshold with conditioning electrical stimuli | During session 1. The estimation of the outcome measurement take approximately 3 minutes.
  The cold detection threshold will be estimated by reducing the temperature until the subjects perceive a cold sensation. Simultaneous will electrical stimulation be applied.
Warm detection threshold | During session 1. The estimation of the outcome measurement take approximately 3 minutes.
  The warm detection threshold will be estimated by increasing the temperature until the subjects perceive a warm sensation.
Warm detection threshold with conditioning electrical stimuli | During session 1. The estimation of the outcome measurement take approximately 3 minutes.
  The warm detection threshold will be estimated by increasing the temperature until the subjects perceive a warm sensation. Simultaneous will electrical stimulation be applied.
Warm pain threshold | During session 1. The estimation of the outcome measurement take approximately 3 minutes.
  The warm pain threshold will be estimated by increasing the temperature until the subjects perceive a painful warm sensation.
Warm pain threshold with conditioning electrical stimuli | During session 1. The estimation of the outcome measurement take approximately 3 minutes.
  The warm pain threshold will be estimated by increasing the temperature until the subjects perceive a warm painful sensation. Simultaneous will electrical stimulation be applied.
Cold pain threshold | During session 1. The estimation of the outcome measurement take approximately 3 minutes.
  The cold pain threshold will be estimated by reducing the temperature until the subjects perceive a painful warm sensation.
Cold pain threshold with conditioning electrical stimuli | During session 1. The estimation of the outcome measurement take approximately 3 minutes.
  The cold pain threshold will be estimated by reducing the temperature until the subjects perceive a cold painful sensation. Simultaneous will electrical stimulation be applied.
The sensation of pulse 1 | During session 1. The estimation of the outcome measurement take approximately 3 minutes.
  The investigator will ask the participant to rate the sensation by a questionnaire. The scale will be 0-10, where 0 indicates no sensation and 10 is the worst imaginable sensation.
The sensation of pulse 2 | During session 1. The estimation of the outcome measurement take approximately 3 minutes.
  The investigater will ask the participant to rate the sensation by a questionnaire. The scale will be from 0-10 where 0 indication no sensation and 10 the worst imaginable sensation.
Perception threshold | During session 1. The estimation of the outcome measurement take approximately 15 minutes.
  The Perception threshold for the cutaneous electrical stimulation will be estimated for two different pulse shapes of the electrical stimulus. The perception threshold is defined as the electrical current needed for the participant to perceive the stimulus. The perception threshold will be estimated by the method of limits.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Tigerholm, Principal Investigator — Aalborg University
Locations (1):
- Aalborg university, Aalborg, North Denmark, Denmark